CLINICAL TRIAL: NCT01733641
Title: Test-Retest Psychometrics of a Novel Neuropsychological Assessment Tool: Reliability Measures for DETECT
Brief Title: Test-Retest Reliability in DETECT
Status: Terminated | Type: Observational
Why Stopped: Limited eligible sample size for study outcomes
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Tamara Espinoza, MD, Instructor, Emory University
Other Study IDs: IRB00052187
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Reliability Properties of a Concussion Screening Tool

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Healthy volunteers without concussion, currently participating in non-or-limited contact sports teams at Emory University will undergo Display Enhanced Testing for Concussion and mild traumatic brain injury (mTBI) (DETECT) on three separate days: at baseline, day 50, and day 90. Prior to enrollment participants will be allocated to the test-retest arm or the exercise arm.

ELIGIBILITY:
Inclusion Criteria:

* age > or = 16
* eligible for active participation during the National Collegiate Athletic Association (NCAA) season or member of the 2011 - 2012 or 2012-2013 club team
* Participation in a non or minimal contact sport

Exclusion Criteria:

* < age 16
* history of concussion in the previous 6 months
* any of the following: learning disabilities, attention deficient disorder, attention deficit hyperactivity disorder, depression or other psychiatric disorder, sleep apnea, seizure disorder, migraine headaches, previous central nervous system (CNS) surgery
* chronic drug or alcohol use; or drug or alcohol use with the previous 24 hours
* inability to complete the study protocol (90 days)

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy volunteer athletes without concussion
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2011-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Primary Objective is to assess the reliability of the DETECT cognitive assessment tool, as measured by changes in DETECT scores from baseline in non-injured athletes. | 90 days
  Subjects will complete the DETECT cognitive assessment tool at Baseline, 50 days, and 90 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Atlanta, Georgia, United States